CLINICAL TRIAL: NCT00085345
Title: Phase II Study of Melphalan, Arsenic Trioxide, and Ascorbic Acid in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: Melphalan, Arsenic Trioxide, and Ascorbic Acid in Treating Patients With Relapsed or Refractory Multiple Myeloma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Oncotherapeutics (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: ONCOTHER-MAC001; CDR0000368637 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2006-07

CONDITIONS: Stage II Multiple Myeloma; Stage III Multiple Myeloma; Refractory Plasma Cell Neoplasm
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Arsenic Trioxide; Ascorbic Acid; Melphalan; Drug Therapy

INTERVENTIONS:
Drug: arsenic trioxide
Drug: ascorbic acid
Drug: melphalan
Procedure: chemosensitization/potentiation
Procedure: chemotherapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as melphalan, arsenic trioxide, and ascorbic acid, work in different ways to stop cancer cells from dividing so they stop growing or die. Arsenic trioxide and ascorbic acid may also help melphalan kill more cancer cells by making them more sensitive to the drugs.

PURPOSE: This phase II trial is studying how well giving melphalan together with arsenic trioxide and ascorbic acid works in treating patients with relapsed or refractory multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the time to progression in patients with relapsed or refractory multiple myeloma (MM) treated with melphalan, arsenic trioxide, and ascorbic acid.
* Determine the response rate (combined complete response, partial response, and minimal response) in patients treated with this regimen.
* Determine the safety and tolerability of this regimen in these patients.

Secondary

* Determine the time to response and overall survival of patients treated with this regimen.
* Determine the effects of this regimen on renal failure associated with MM in these patients.

OUTLINE: This is an open-label, non-randomized, multicenter study.

Patients receive oral melphalan once daily on days 1-4 of week 1 and arsenic trioxide (ATO) IV over 1-2 hours and ascorbic acid IV over 15 minutes on days 1-4 of week 1 and then twice weekly during weeks 2-5. Treatment repeats every 6 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients with disease progression any time after course 1 also receive oral prednisone once daily on days 1-4 and 22-25 of each course. Patients achieving a complete response after 6 courses of therapy undergo bone marrow biopsy and receive no further therapy. Patients achieving stable disease or a partial response after 6 courses of therapy continue to receive ATO and ascorbic acid once weekly.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 65 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of multiple myeloma meeting at least 1 of the following criteria:
* Relapsed disease after a response to standard first-line chemotherapy (e.g., vincristine, doxorubicin, and dexamethasone [VAD] OR melphalan and prednisone) or first-line high-dose chemotherapy
* Refractory disease (failed to achieve at least stable disease) to most recent chemotherapy with or without systemic corticosteroids
* Measurable disease, defined as a monoclonal immunoglobulin spike on serum electrophoresis of ≥ 1 g/dL AND/OR urine monoclonal immunoglobulin spike of ≥ 200 mg/24 hours
* No non-secretory myeloma
* No plasma cell leukemia

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 60-100%

Life expectancy

* More than 3 months

Hematopoietic

* Platelet count ≥ 50,000/mm^3 (30,000/mm^3 if bone marrow is extensively infiltrated)
* Hemoglobin ≥ 8.0 g/dL
* Absolute neutrophil count ≥ 1,000/mm^3
* Pancytopenia secondary to multiple myeloma or hypersplenism allowed

Hepatic

* AST and ALT ≤ 3 times upper limit of normal (ULN)
* Bilirubin ≤ 2 times ULN (unless clearly related to disease)
* No known active hepatitis B or C infection

Renal

* Calcium < 14 mg/dL

Cardiovascular

* No evidence of acute ischemia or new conduction system abnormality by electrocardiogram
* No myocardial infarction within the past 6 months
* No New York Heart Association class III or IV heart failure
* No poorly controlled hypertension
* No prolonged corrected QT interval (> 460 ms) with potassium > 4 mmol/L and magnesium ≥ 1.8 mmol/L

Other

* No active infection
* No POEMS syndrome (plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes)
* No diabetes mellitus
* No other serious medical or psychiatric illness that would preclude study participation
* No known allergic reaction attributable to compounds of similar chemical or biological composition to study drugs
* No history of grand mal seizures
* HIV negative
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 4 weeks since prior immunotherapy or antibody therapy

Chemotherapy

* See Disease Characteristics
* More than 3 weeks since prior chemotherapy (6 weeks for nitrosoureas)

Endocrine therapy

* See Disease Characteristics
* No other concurrent corticosteroids

Radiotherapy

* More than 4 weeks since prior radiotherapy

Surgery

* More than 4 weeks since prior major surgery

Other

* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James R. Berenson, MD, Study Chair — Oncotherapeutics
Locations (19):
- United States (19):
  - Palo Verde Hematology Oncology, Glendale, Arizona
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - Southbay Oncology / Hematology Medical Group, Campbell, California
  - Fountain Valley, California
  - Hematology-Oncology Medical Group of Fresno, Incorporated, Fresno, California
  - Hematology Oncology Medical Group of Orange County, Incorporated, Orange, California
  - Cancer Care Associates Medical Group - Redondo Beach, Redondo Beach, California
  - Redwood Regional Oncology Center - Sotoyome, Santa Rosa, California
  - Cancer Prevention and Treatment Center at Dominican and Watsonville Community Hospital, Soquel, California
  - San Diego Cancer Center - Vista, Vista, California
  - Oncotherapeutics, West Hollywood, California
  - Mount Sinai Comprehensive Cancer Center at Mount Sinai Medical Center, Miami Beach, Florida
  - Atlanta Cancer Care - Roswell, Roswell, Georgia
  - Tulane Cancer Center at Tulane University Hospital and Clinic, New Orleans, Louisiana
  - Center for Cancer and Blood Disorders at Suburban Hospital, Bethesda, Maryland
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Hackensack University Medical Center Cancer Center, Hackensack, New Jersey
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Utah Cancer Specialists - Administrative Office, Salt Lake City, Utah